CLINICAL TRIAL: NCT03685188
Title: Comparison of Oxycodone and Sufentanil for Analgesic Efficacy After Hip Surgery: a Prospective, Multicenter Randomized Controlled Trial
Brief Title: Oxycodone and Sufentanil for Analgesia in Hip Surgery
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Associate professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCH2018086
Record Dates: First submitted 2018-09-13; First posted 2018-09-26 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Analgesia, Patient-Controlled
Keywords: Randomized controlled trial; oxycodone; sufentanil; patient-controlled intravenous analgesia; hip surgery
MeSH Terms: conditions — Agnosia | interventions — Oxycodone; Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxycodone group (Experimental): PCIA is formulated at 0.4 mg/ml of oxycodone.
  Interventions: Drug: Oxycodone Hydrochloride
- Sufentanil group (Active Comparator): PCIA is formulated at 2 μg/ml of sufentanil.
  Interventions: Drug: Sufentanil Citrate

INTERVENTIONS:
Drug: Oxycodone Hydrochloride — Subjects will receive patient' controlled intravenous analgesia in analgesic pump with 0.4 mg/ml of oxycodone for postoperative analgesia.
  Arms: Oxycodone group
Drug: Sufentanil Citrate — Subjects will receive patient' controlled intravenous analgesia in analgesic pump with 2 μg/ml of sufentanil for postoperative analgesia.
  Arms: Sufentanil group

SUMMARY:
We design this randomized controlled trial to compare the safety and efficacy of Oxycodone and Sufentanil for postoperative patient-controlled analgesia in patients undergoing hip surgery, with a view to finding the optimal postoperative analgesic regime with fewer adverse reactions and promoting patients' rehabilitation.

DETAILED DESCRIPTION:
Hip surgery is a common type of orthopedic surgery. The pathologies are complex, including chronic conditions such as femoral head necrosis, primary hip dysplasia, hip joint osteoarthritis and rheumatoid arthritis, as well as acute diseases such as femoral neck fractures and intertrochanteric fractures. The surgical treatment includes closed reduction and internal fixation, open reduction and internal fixation, hemiarthroplasty (femoral head replacement), and total hip arthroplasty, etc. The population of patients undergoing hip surgery has a high proportion of elderly (>65 years old), with multiple preoperative comorbidities, and significant postoperative pain. We must achieve the balance between the providing sufficient analgesia and minimizing associated adverse reactions perioperatively for such group of patients, therefore promoting patients' rehabilitation.

Sufentanil, a pure μ receptor agonist with active metabolite, is a long-acting strong opioid which has high analgesic efficacy. It is commonly used in anesthesia practice, not only for intraoperative analgesia, but also postoperative pain relief, i.e. a popular drug of choice used for Patient Control Intravenous Analgesia (PCIA). However, sufentanil is associated with high incidence of postoperative nausea and vomiting (PONV), respiratory depression and other adverse reactions, which could negatively affect the patient's analgesic satisfaction, and compromise the course of postoperative recovery. It is important to establish an effective and safe postoperative analgesic regime that can achieve the comparable analgesic efficacy with reduced incidence of adverse reactions. Oxycodone is a semi-synthetic opioid which is extracted from the thebaine, it activates both μ and κ opioid receptors. It has been reported to have good analgesic effect and lower incidence of adverse reactions such as PONV in comparison with Morphine, and could be a reasonable option for PCIA. As Oxycodone can agonize κ receptors and reduce visceral pain, most of the existing studies on Oxycodone are focused on laparoscopic cholecystectomy and other abdominal surgeries, with the average age of study patients is between 40 to 55 years old, and also lack of large sample studies.

Based on the abovementioned literatures, we propose the hypothesis that in hip surgery, compared with Sufentanil PCIA, the equipotency dose of Oxycodone PCIA can achieve the same postoperative analgesic efficacy and may also reduce the incidence of adverse reactions associated with opioids.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing unilateral hip surgery, sign the "informed consent form".
* Age above 18 years old, with both genders.

Exclusion criteria:

* Pregnant or lactating women.
* Patient with history of drug abuse, including but not limited to opioids, amphetamines, ketamine, etc.
* Allergic to opioids or any other anesthetic agent.
* History or family history of malignant hyperthermia.
* Have history of nervous system diseases such as peripheral neuropathy, psychiatric mental illness, or postoperative delirium.
* Other conditions that the investigators consider unsuitable for participation in the study, such as Parkinson's disease, unable to communicate, or impairment of cognitive function etc.
* Participation in another trial in the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative numerical rating scales (NRS) at rest | Up to 72 hours after operation
  Resting NRS pain scores at 2 h after surgery.

SECONDARY OUTCOMES:
Incidence of post operative nausea and vomiting (PONV) | Up to 72 hours after operation
  The proportion of subjects who experienced PONV
The severity of first PONV and the most severe PONV | Up to 30 days after operation
  The severity of PONV is scored from 0 to 10, and 0 represents no PONV at all, and 10 represents very severe PONV.
Time from the end of operation to the first onset of PONV | Up to 30 days after operation
  Time from the end of operation to the first onset of PONV
Postoperative numerical rating scales (NRS) at rest | Up to 72 hours after operation
  Postoperative resting NRS pain scores at 30 min, 6h, 24h, 48h, and 72h after the surgery
Postoperative NRS on movement | Up to 72 hours after operation
  Postoperative NRS pain score on movement, up to 72hr.
Postoperative complications | Up to 30 days after operation
  Incidence of postoperative adverse reactions and complications, which are divided into five grades:
  1. Grade Ⅰ ： Recovery after temporary treatment, e.g., postoperative anxiety, insomnia.
  2. Grade Ⅱ ： Prolonged hospitalization, e.g., pulmonary infection requiring antibiotics or other treatment, surgical wound infection requiring wound deb-ridement.
  3. Grade Ⅲ： Life threatening complications requiring intense treatment dur-ing hospitalization, and resulting in good functional recovery e.g., dialysis thera-py for acute renal insufficiency, mechanical ventilatory support for respiratory failure, or postoperative bleeding requiring re-operation.
  4. Grade Ⅳ： Life threatening complications resulting in significantly de-creased quality of life, e.g., myocardial infarction, stroke that left with paralytic limbs.
  5. Grade Ⅴ： All-cause mortality by 30 days after operation.
Motion of hip joints | Up to 72 hours after operation
  Range of motion of hip joints during 3 days after operation.
Straight leg raising time | Up to 72 hours after operation
  Time from the end of operation to the time that patient can raise his affected lower limb by himself (Unit: hour).
Ground exercise time | Up to 72 hours after operation
  Time from the end of operation to the time that patient can do the ground exercise by himself (Unit: hour).
Mobilization time | Up to 72 hours after operation
  Time frame from the end of operation to able to walk without external assistance (Walking aids such as crutches can be used, unit: hour).
Residual amount of drug | Up to 72 hours after operation
  Residual amount of drug in the analgesic pump.
Postoperative analgesics requirement | Up to 72 hours after operation
  Postoperative analgesics requirement during 3 days after operation
Total in-hospital cost. | Up to 30 days after operation
  Total hospitalization expenses after the destruction of costly consumables in orthopedic operation.
Length of stay (LOS) in hospital | Up to 30 days after operation
  Time frame from the day of hospital admission to discharge from the hospital (unit: days)
Postoperative LOS | Up to 30 days after operation
  Time frame from the day of operation to discharge from the hospital (unit: days).
Re-admission rate | Up to 30 days after operation
  The incidence of re-admission within 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liao C, Zhu H, Zhong J, Lai X, Zhang B, Liao R. Patient Controlled Intravenous Analgesia with Oxycodone or Sufentanil After Hip Surgery: Study Protocol for a Multi-Centered, Randomized Controlled Trial. J Clin Med. 2025 Feb 25;14(5):1525. doi: 10.3390/jcm14051525. PMID 40095065